CLINICAL TRIAL: NCT04011904
Title: The Role of Traditional or Western Diet in the TBC1D4 Gene on Glucose
Brief Title: The Role of Traditional or Western Diet in the TBC1D4 Gene on Glucose Homeostasis in Greenland Inuits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Professor Lotte Lauritzen, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: KVUG 2018-26
Record Dates: First submitted 2019-05-13; First posted 2019-07-09 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: T2D
Keywords: Greenland Inuit; Traditional diet; TBC1D4
MeSH Terms: interventions — Cross-Over Studies

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Inuit Diet (Experimental): This will be a traditional Inuit diet (TID) rich in marine mammals (such as walrus, seal, and whale), fish, caribou and musk ox, with low intake of grains, fast food and other imported foods. The TID diet will be high in fat (>40 of the energy (E%)) and low in carbohydrate (<30 E%).
  Interventions: Other: Cross-over study
- Westernized Diet (Placebo Comparator): This will be a Westernized diet will be consisting of high amounts of grains, potatoes, rice and imported meats from livestock animals (beef, pork and chicken). The Westernized diet will be high in carbohydrate (55-65 E%) and lower in fat (30-35 E%).
  Interventions: Other: Cross-over study

INTERVENTIONS:
Other: Cross-over study — Traditional Inuit Diet vs Westernized Diet

SUMMARY:
Studies of Greenland Inuit before the 1980s found a low prevalence of type 2 diabetes (T2D) compared to Western populations. However, recent population studies in Greenland found a notably high prevalence of diabetes (9%) and pre-diabetes (19%) in the adult population.

In many studies worldwide an increase in obesity, diabetes, and cardiovascular disease has been ascribed to social transition and in particular urbanization, but the Inuit in Greenland do not fit the pattern. Paradoxically, the highest prevalence of diabetes is seen in the least urbanized areas. Thus, while previously rare, T2D has become epidemic in Inuit. In a recent study by Moltke et al found that a variant in the TBC1D4 gene was strongly associated with insulin resistance in skeletal muscle, high postprandial blood glucose and a high risk of T2D.

The rapid increase in the prevalence of T2D and other metabolic traits and the well documented genetic susceptibility indicates that lifestyle components, particularly physical activity, and diet significantly modify the genetic effects on glucose homeostasis. Thus, changing dietary habits from a diet high in traditional foods, mostly consisting of marine mammals and fish (high in protein and unsaturated fats, and low in carbohydrate) to a westernized diet, with high contents of sugar and saturated fat may have increased the T2D incidence in Arctic Inuit.

The investigators will perform a 4-week cross-over intervention study of the traditional diet versus a western diet among homozygous carriers and WTs on 2-hour glucose after an oral glucose tolerance test (OGTT). In addition, the investigators will examine the effects on cardiometabolic abnormalities such as low-grade systemic inflammation and dyslipidemia. Furthermore, the investigators will characterize the metabolic phenotype of participants, as well as gut microbiota and brown adipose tissue markers to elucidate the molecular mechanisms underlying potential improvements of a traditional Inuit diet.

DETAILED DESCRIPTION:
The overall objective of the study is to investigate whether a traditional marine diet high in fat and low in carbohydrate compared to a westernized diet could improve glycemic control in Greenland Inuit. Furthermore, the objective is to study whether the genetic risk of postprandial hyperglycemia among Greenlandic carriers of the common nonsense p.Arg684Ter variant in the TBC1D4 gene is modified to a larger degree by the diet compared to non-carriers.

The investigators will perform a 4-week cross-over intervention study of the traditional diet versus a western diet among homozygous carriers and WTs on 2-hour glucose after an oral glucose tolerance test (OGTT). In addition, the investigators will examine the effects on cardiometabolic abnormalities such as low-grade systemic inflammation and dyslipidemia. Furthermore, the investigators will characterize the metabolic phenotype of participants, as well as gut microbiota and brown adipose tissue markers to elucidate the molecular mechanisms underlying potential improvements of a traditional Inuit diet.

The study is expected to provide relevant information in relation to whether diet has a role in preventing T2D in the large group of people who are hetero / homozygous for the TBC1D4 variant. The investigators expect this enhanced insight to be useful and valuable for future development of genotype based interventions for these persons.

For the individual participant, the results of the study are expected to provide constructive knowledge to guide the participants in which actions they could take to reduce the likelihood of developing T2D.

Hypothesis

The investigators hypothesize that the traditional marine diet very high in fat and low in carbohydrates will improve postprandial glucose handling in Greenland Inuit. Furthermore, the investigators hypothesise that this effect is modified among carriers of the common nonsense p.Arg684Ter variant in the TBC1D4 gene which will have larger effects of following the traditional marine diet.

Methodology

Overall study design 30 homozygous carriers and 30 homozygous non-carriers of the nonsense p.Arg684Ter variant in the TBC1D4 gene between 18-80 years will be included in the study.

The study will be conducted as a randomized, controlled, cross-over design, comprising two dietary intervention periods of four weeks duration, with no washout in between. The participants will be randomized to start on one of the two diet periods and cross-over to the other dietary period at 4 weeks (see figure 1). The investigators expect to recruit participants after approval from April 2019 and have the last patient last visit by September 2020. Recruitment of study participants will be based on the currently ongoing Greenland Population Study (project 2017-5582) to ensure that the investigators have 50% homozygous carriers of the nonsense p.Arg684Ter variant in the TBC1D4 gene. The study will be carried out in three geographical areas: Nuuk, Qaanaaq, and Qasigiannguit.

Randomization, allocation, concealment, and blinding

After having given oral and written consent, randomization will be performed separately for each participant based on the genotype in blocks of variable size to ensure equal randomization throughout the enrolment phase of the study. The randomization sequence will be done by an investigator without contact to the participants. The personnel conducting the study will allocate participants to the sequence of intervention using a list of participant IDs matched with allocated sequences. Blinding participants is not feasible due to the nature of the intervention, however blinding of the allocation sequence will be established during sample analysis and initial data analysis.

Intervention

Two diets will be designed for the intervention. A traditional Inuit diet (TID) rich in marine mammals (such as walrus, seal, and whale), fish, caribou and musk ox, with low intake of grains, fast food, and other imported foods. The TID diet will be high in fat (>40 of the energy (E%)) and low in carbohydrate (<30 E%). The Westernized diet will be consisting of high amounts of grains, potatoes, rice and imported meats from livestock animals (beef, pork, and chicken). The Westernized diet will be high in carbohydrate (55-65 E%) and lower in fat (30-35 E%). Major parts (20-25E%) of the diet will be given to the participants upon start and during the study in the form of frozen goods. For the TID group, this will be marine mammals and fish, while for the Westernized group the products delivered will mainly be grains and livestock animals. Instructions for the participants regarding the incorporation of dietary changes will be performed by trained study staff.

Study products

Assessment of habitual food intake at baseline will be conducted with a previously validated food frequency questionnaire. A modified version of the food frequency questionnaire will be used at the end of each intervention period for assessing habitual diet during the intervention period. In addition, participants will be asked to keep a simple log of ingestion of delivered products to estimate compliance. The investigators will apply for sponsorship for study products. The potential study product sponsors will play no role in the design, methods, data management and analysis or in the decision to publish.

Consumption of Study products

Trained study personnel will provide participants with instructions on how to incorporate the provided study products in the diet. Initially, it will be ensured that the study products are provided in sufficient amounts to ensure ad libitum consumption. Participants will be provided individualized amounts of all study products every second week. All study products are provided as fresh or frozen products, and all food products will be picked up at the local study site.

Study examinations

Participants will arrive for clinical examination after an overnight fast of at least 8 hours. Lifestyle questionnaires, including a food frequency questionnaire and questionnaires about medication use, will be performed for baseline characterization of the participants. Blood pressure and anthropometric measurements are performed including measurements of body weight, height, waist and hip circumference, sagittal abdominal diameter and bio-impedance measurements for assessing body fat mass. A fasting blood sample is obtained and an OGTT is performed with collection of blood samples after 0, 30 and 120 min. Samples will be analyzed with standard clinical procedures for glycaemic variability markers, including glucose, insulin, c-peptide, and HbA1c, as well as plasma lipids. Circulating fatty acids profiles will be used as a marker of compliance with the TID using dried blood spots. Furthermore, fecal samples will be collected at all examination visits and kept stored for future microbiota analyses, using untargeted shotgun sequencing. Biobanked samples will be stored for further analyses which could include gastrointestinal hormones, gut microbiota metabolites, additional compliance markers such as alkylresorcinols (for grain intake) low-grade inflammation markers and markers of brown fat accumulation. In addition, participants will be equipped with a 24-h continuous glucose monitoring device for 14 days at the end of each intervention period. All 3 examination days consists of similar examinations and data collections and are estimated to last approximately 5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided written informed consent
* Age between 18 and 80 years
* Homozygous carriers of the nonsense p.Arg684Ter variant in the TBC1D4 gene (cases)
* Homozygous non-carriers of the nonsense p.Arg684Ter variant in the TBC1D4 gene (control)

Exclusion Criteria:

* If study participants do not want to know whether they are carriers or non-carriers of the p.Arg684Ter variant in the TBC1D4 gene they will not be able to participate in the study
* BMI ≥ 18.5 kg/m2
* Diagnosis of diabetes (HbA1c ≥ 6,5% (48 mmol/mol)) or pharmacological treatment of diabetes (10).
* Use of peroral glucocorticoids
* Lack of compliance with the procedures in the study protocol, judged by Investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Changes in 2-h post-OGTT glucose in blood between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  2 hour post oral glucose tolerance test glucose mesurement in blood (mmol/L)

SECONDARY OUTCOMES:
Changes in Hba1c between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  fasting measurement of blood glycated hemoglobin (%)
Changes in fasting blood glucose between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  Fasting measurement of blood glucose (mmol/L)
Changes in 30 min post OGTT between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  Measurement of blood glucose 30 min after OGTT (mmol/L)
Continuous glucose monitoring | Week 2 and Week 6
  Continuous glucose monitor from Abbott is worn for 14 days in each period providing glucose measurements continuously (mmol/L).
Insulin sensitivity and secretion | Week 1, Week 4 and week 8
  Measured as part of the OGTT. Plasma glucose (mmol/l). Plasma insulin - fasting (pmol/l)
Changes in blood lipids between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  Measurements of total and HDL cholesterol (mmol/L) and triglycerides (mmol/L).
Changes in gastrointestinal hormones between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  Measurements of e.g. GLP-1, PYY and GIP (pmol/L) in blood.
Changes in gut microbiota composition between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  Measured on fecal samples
Changes in C-Reactive Protein between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  Blood measurements of C-Reactive Protein (mg/L)
Changes in Interleukin-6 between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  Blood measurements of Interleukin-6 (pg/mL)
Changes in small metabolites between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  Measured using blood metabolomic measurements of amino acids, lipids, and other small metabolites (umol/L)
Changes in weight between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  Measured using a Tanita body composition analyser. Body weight in kilograms
Changes in body composition between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  Measured using a Tanita body composition analyser. Fat free mass and Body fat mass in kilograms used to calculate body fat percentage.
Changes in waist and hip circumference between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  Measured using measurement tape
Changes in fatty acids (compliance measurement) between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  Objective measures of compliance with fish intake, fatty acids (%FA) in blood.
Changes in alkylresorcinols (compliance measurement) between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  Objective measures of compliance with grain intake, alkylresorcinols (umol/L) in blood.
Changes in blood pressure (BP) between the baseline and endpoint change in the two periods | Week 1, Week 4 and week 8
  Systolic BP (mmHG) Diastolic BP (mmHG)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Exercise, Nutrition and Sports, Faculty of Sciences, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moller G, Lind MV, Hauptmann AL, Senftleber N, Hansen CB, Hansen T, Jorgensen ME, Lauritzen L. The role of a traditional and western diet on glucose homeostasis in Greenlandic Inuit carriers and non-carriers of type 2 diabetes variant in the TBC1D4 gene: A protocol for a randomized clinical trial. Contemp Clin Trials Commun. 2021 Jan 27;21:100734. doi: 10.1016/j.conctc.2021.100734. eCollection 2021 Mar. PMID 33604488